CLINICAL TRIAL: NCT00538967
Title: The Effect of Doxycycline on Matrix Metalloproteinase Expression and Activity in the Abdominal Aneurysm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P00.146
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-10

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Collagenases; MMP; Cathepsins; Doxycycline; Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (No Intervention)
- 2 (Active Comparator): doxycycline 50 mg/day
  Interventions: Drug: doxycycline
- 3 (Active Comparator): doxycycline 100 mg
  Interventions: Drug: doxycycline
- 4 (Active Comparator): doxycycline 300 mg
  Interventions: Drug: doxycycline

INTERVENTIONS:
Drug: doxycycline — 2 weeks once daily
  Arms: 2; 3; 4

SUMMARY:
The matrix metalloproteinase-9 (MMP-9) is considered to play a central role in abdominal aortic aneurysm (AAA) initiation. Doxycycline has direct MMP-9 inhibiting properties in vitro, and it effectively suppresses AAA development in rodents. Observed inhibition of AAA progression, and contradictory findings in human studies evaluating the effect of doxycycline therapy on aortic wall MMP-9 suggest that the effects of doxycycline extend beyond MMP-9 inhibition, and that the effect may be dose dependent.

DETAILED DESCRIPTION:
In this clinical trial, we evaluated the effect of two weeks of low (50 mg/day), medium (100 mg/day) or high dose (300 mg/day) doxycycline versus no medication in patients undergoing elective AAA repair. The effect of doxycycline treatment on MMP and cysteine proteases, and their respective inhibitors was evaluated in an integrative approach.

ELIGIBILITY:
Inclusion Criteria:

* Elective open aneurysm repair

Exclusion Criteria:

* Severe kidney and liver dysfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2002-05; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Collagenase mRNA and protein expression | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jan HN Lindeman, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands